CLINICAL TRIAL: NCT04040920
Title: The Effect of Ozone Application Before Fissure Sealants: a Split Mouth Randomized Controlled Trial
Brief Title: Ozone Application Before Fissure Sealants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC 02/2019
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Caries,Dental
Keywords: Ozone; Pits and fissures sealants; Prevention
MeSH Terms: conditions — Dental Caries | interventions — Pit and Fissure Sealants

STUDY DESIGN:
Intervention Model Description: Splith mouth design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ozone therapy (Experimental): Ozone application before pits and fissure sealants
  Interventions: Device: Ozone; Other: Pits and fissure sealants
- Pits and fissure sealants (Active Comparator)
  Interventions: Other: Pits and fissure sealants

INTERVENTIONS:
Device: Ozone — One minute of pretreatment with ozone by using the OzoneDTA device
  Arms: Ozone therapy
Other: Pits and fissure sealants — cleansing of the occlusal surfaces with a nylon brush and polishing toothpaste; surface etching with 36% orthophosphoric acid for 30'', surface cleaning and drying for 30 '', application of the sealing material, polymerization for 60'';

SUMMARY:
Decay is a multifactorial infective degenerative disease of hard dental tissues, caused by Streptococcus mutans and Lactobacillus forming the bacterial biofilm of teeth surfaces. Decays generally evolve in fissures and pits of secondary molars. Pits and fissure sealants prevent decays if performed in two years from eruption. Ozone has bactericidal effect and remineralizing capacity on enamel.

The aim of this study is to assess the effectiveness of ozone application before sealants in increasing their duration in time.

ELIGIBILITY:
Inclusion Criteria:

* first or second secondary molars to be sealed
* possibility to isolate with rubber dam both the teeth involved
* no clear signs of pigmentations
* good general health

Exclusion Criteria:

* latex allergy
* epilepsy or other severe neurological pathologies
* psychiatric disease
* excessive sensibility to electrical current
* severe asthma
* enamel disorders, such as amelogenesis imperfect, white spots, fluorosis or Molar Incisors Hypomineralization

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sealants failure | 12 months after sealant
  Frequency of sealed failure defined as presence of to one or more of these outcomes: Marginal fissure; Sealant fracture; Decay; Marginal pigmentations; Sealant detachment Evaluation of the relative frequency of the different causes of failure

SECONDARY OUTCOMES:
Sealants failure | 6 months after sealant
  Frequency of sealed failure defined as presence of to one or more of these outcomes: Marginal fissure; Sealant fracture; Decay; Marginal pigmentations; Sealant detachment Evaluation of the relative frequency of the different causes of failure
Sealants failure | 24 months after sealant
  Frequency of sealed failure defined as presence of to one or more of these outcomes: Marginal fissure; Sealant fracture; Decay; Marginal pigmentations; Sealant detachment Evaluation of the relative frequency of the different causes of failure
Secondary decay in failed sealants | 6 months after sealant
  Frequency of secondary decay in teeth with failed sealants
Secondary decay in failed sealants | 12 months after sealant
  Frequency of secondary decay in teeth with failed sealants
Secondary decay in failed sealants | 24 months after sealant
  Frequency of secondary decay in teeth with failed sealants

CONTACTS AND LOCATIONS:
Overall Officials: Milena Cadenaro, DDS,MSc,PhD, Study Chair — IRCCS Burlo Garofolo; Maddalena Chermetz, DDS,MSc, Principal Investigator — IRCCS Burlo Garofolo
Locations (1):
- Institute for Maternal and Child Health - IRCCS Burlo Garofolo-, Trieste, Trieste, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data collected during the study will be available from the Study Director on reasonable request after evaluation of a protocol approved by an Ethical Committee
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of data on peer reviewed journals
Access Criteria: Data collected during the study will be available from the Study Director on reasonable request after evaluation of a protocol approved by an Ethical Committee